CLINICAL TRIAL: NCT01523106
Title: L-carnitine to Treat Fatigue Associated With Crohn's Disease
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: carnitine and crohn's disease
Record Dates: First submitted 2012-01-18; First posted 2012-02-01 (Estimated); Last update posted 2014-01-17 (Estimated); Status verified 2014-01

CONDITIONS: Crohn's Disease; Fatigue
Keywords: Crohn's disease; carnitine
MeSH Terms: conditions — Crohn Disease; Fatigue | interventions — Carnitine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Carnitine (Active Comparator): Patients will take 4grams of L-carnitine (2 grams twice daily) for 3 months
  Interventions: Drug: L-carnitine
- Placebo (Placebo Comparator): Patients will take placebo for 3 months. Placebo is manufactured by the same company as the L-carnitine and will have a similar appearance.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: L-carnitine — dietary supplement
  Arms: Carnitine
Other: Placebo — Patients will receive placebo, which will be manufactured by the same supplier as L-carnitine and appears identical. Patients will take an equal number of pills (8 pills/day).
  Arms: Placebo

SUMMARY:
This is a randomized, double-blind, placebo-controlled study, comparing the effect of L-carnitine vs placebo on fatigue among Crohn's disease patients.

The specific aim of this study is to determine if treatment with L-carnitine is more effective than placebo at decreasing fatigue severity scores, while accounting for disease activity and concomitant anemia, depression/anxiety and poor sleep quality.

DETAILED DESCRIPTION:
A total of 100 patients will be recruited, in order to be able ensure to detect a significant difference in fatigue between the treatment and control groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients will have had previously macro- and microscopically verified Crohn's disease, as defined by traditional clinical and endoscopic standards.
* To be included, patients need to have disease which is either in remission or is mild to moderate in severity, as defined by the Harvey-Bradshaw Index Score (HBI<16).
* In addition, patients will need to answer "yes" to the screening study entry question ("Is fatigue a signficant problem for you currently?").

Exclusion Criteria:

* Exclusion criteria will include:

  * age <18 or >70 years
  * pregnancy or delivery within 6 months
  * malignancy diagnosed within 1 year
  * oral/intravenous steroid treatment within 6 months
  * any surgery within 6 months
  * presence of a stoma or ileo-anal J-pouch anastomosis
  * concurrent hepatitis B or C infection
  * cirrhosis
  * renal insufficiency (CrCl<60) and history of seizure disorder or hypothyrodism.
  * prior to study enrollment
  * women of child-bearing age will need to undergo pregnancy testing.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-08; Primary Completion 2014-02 (Estimated); Study Completion 2014-02 (Estimated)

PRIMARY OUTCOMES:
Change in fatigue severity scale | From baseline to 3 months after intervention initiation
  The Fatigue Severity Score is a validated instrument to assess fatigue associated with chronic disease. The scale ranges from scores from 9 to 63, with a higher score indicated greater fatigue.

SECONDARY OUTCOMES:
Change in Multidimensional Fatigue Inventory | From baseline to 3 months after intevention initiation
  This is a validated instrument to measure fatigue and has been validated for use for patients with inflammatory bowel disease. Scores range from 4-20, with higher scores indicated more severe fatigue.
Change in handgrip strength | From baseline to 3 months after treatment intervention
  Handgrip strength will be assessed by a portable dynanometer. Maximal force after three tries will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Uma Mahadevan, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF Medical Center, Mt. Zion Medical Center, San Francisco, California, United States